CLINICAL TRIAL: NCT03187561
Title: Coparenting, Infant Sleep, and Infant Development
Acronym: SIESTA-FF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Penn State University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Douglas M. Teti, Professor of HDFS, Psychology, and Pediatrics, Penn State University
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: STUDY00006724; R01HD088566 (NIH)
Record Dates: First submitted 2017-06-09; First posted 2017-06-15 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Sleep; Parenting; Marital Relationship; Parent-Child Relations
Keywords: Sleep; Parenting; Marital relationship; Parent-child relations

STUDY DESIGN:
Intervention Model Description: In the proposed 3-arm RCT, in one arm families will experience Family Foundations (FF) intervention as originally formulated; in the second, families will receive an adapted FF (FF+) program that emphasizes coparenting in infant sleep contexts; the third arm will serve as controls.
Who Masked: Participant, Outcomes Assessor
Masking Description: All participants will be informed that they are being recruited into an intervention study targeting coparenting, but participants will not be informed about which arm of the study to which they have been assigned. Data collectors and outcome assessors will not be informed about which arm of the study to which participants have been assigned, to assure that all outcomes and evaluations of intervention are conducted blindly, to avoid experimenter bias.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Family Foundations (FF) (Experimental): The original Family Foundations transition-to-parenthood coparenting intervention will be implemented to all participants assigned to this arm
  Interventions: Behavioral: Infant sleep-adapted coparenting intervention
- Sleep-adapted Family Foundations (FF+) (Experimental): A sleep-adapted Family Foundations transition-to-parenthood coparenting intervention will be implemented to all participants in this arm. The adaptation will be an emphasis on coparenting in relation to infant sleep concerns and activities.
  Interventions: Behavioral: Infant sleep-adapted coparenting intervention
- Control (Other): Participants in this arm will not receive either intervention.
  Interventions: Behavioral: Infant sleep-adapted coparenting intervention

INTERVENTIONS:
Behavioral: Infant sleep-adapted coparenting intervention — The Family Foundations intervention, as originally formulated, and a sleep-adapted Family Foundations intervention, will be implemented to participants in arm 1 and arm 2, respectively.

SUMMARY:
This 3-arm RCT tests the effects of a sleep-enhanced adaptation (FF+) of a well-known, evidence-based transition-to-parenting coparenting intervention program (Family Foundations; FF). In one arm, families will experience FF as originally formulated; in the second, families will receive an adapted FF (FF+) program that emphasizes coparenting in infant sleep contexts; the third arm will serve as controls. It is hypothesized that (1) Compared to controls, parents in both FF groups will report improved overall coparenting and reduced overall distress, but parents in the FF+ group will show greater improvements in coparenting and individual parenting in infant sleep contexts, better infant and parent sleep, and better child adjustment; (2) early coparenting around infant sleep will be a central mechanism by which both interventions exert their effects.

DETAILED DESCRIPTION:
Although infant sleep regulation across the first year proceeds well for many infants, for many infants that is not the case, and estimates of sleep problems among infants and preschoolers range between 25%-33%. Dysregulated infant sleep is predictive of poor parent sleep, and chronic sleep disruption can place families in turmoil, with consequences for the marital and coparenting relationship. Further, mothers reporting early coparenting distress are at risk for personal distress and poor bedtime and nighttime parenting, which in turn predicts infant sleep problems and insecure infant attachment. This application proposes a randomized clinical trial (RCT) to evaluate the effects of a sleep-enhanced adaptation of an evidence-based transition-to-parenting coparenting intervention program [Family Foundations - FF). The rationale for this study is twofold. First, recent findings from the PI's Project SIESTA (R01HD052809) indicate that poor coparenting at one month post-partum predicts persistent infant-parent co-sleeping across the first year, elevated maternal depressive symptoms, emotionally unavailable bedtime parenting, and insecure infant-mother attachments. Second, whereas FF as originally developed has been successful in improving coparenting, marital adjustment, and overall parenting quality, it gives little specific attention to coparenting in infant sleep contexts, which SIESTA findings identify as critically important to parent and infant outcomes later in the first year. The proposed 3-arm RCT responds to these concerns. In one arm, families will experience FF as originally formulated; in the second, families will receive an adapted FF that emphasizes coparenting in infant sleep contexts; the third arm will serve as controls. Assessments of coparenting and parenting in infant sleep contexts, parental adjustment to infant sleep behavior, choices about sleep arrangements, infant and parent sleep quality, and infant socio-emotional functioning, will serve as outcomes. Our central hypotheses are: (1) Compared to controls, parents in both FF groups will report improved overall coparenting and reduced overall distress, but parents in the adapted FF group will show greater improvements in coparenting and individual parenting in infant sleep contexts, better infant and parent sleep, and better child adjustment; (2) early coparenting around infant sleep will be a central mechanism by which both interventions exert their effects. This research is foundational to a broader understanding of coparenting processes that underlie successful family transitions and contributes to the refinement of a successful coparenting program. Study results will be of immediate use to obstetric and pediatric services interested in augmenting childbirth education material with information on coparenting practices in infant sleep contexts.

ELIGIBILITY:
Inclusion Criteria:

* Two-parent families (married or living with a partner
* Families pregnant with their first child, of any race/ethnicity
* Parents who can understand and speak English
* Parents over the age of 18
* Parents living in independent units

Exclusion Criteria:

* Single-parent families
* Families pregnant with a second born or later born child
* Families who cannot speak and understand English
* Families in which one parent under the age of 18
* Parents living with families of origin

Ages: 1 Month to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 216 (Actual)
Dates: Start 2018-11-15 (Actual); Primary Completion 2025-05-09 (Actual); Study Completion 2025-05-09 (Actual)

PRIMARY OUTCOMES:
Overall coparenting quality | 12 months post-partum
  Quality of coparenting
Quality of coparenting around infant sleep contexts | 1 month post-partum
  Quality of coparenting regarding decisions parents make about infant sleep
Quality of infant sleep | 6 months post-partum
  Infant sleep quality from actigraphy and infant sleep diaries reported by parents
Quality of parent sleep | 6 months post-partum
  Sleep quality for each parent, from actigraphy and sleep diary information
Attachment Q-Set | 12 months post-partum
  Quality of infant attachment to mother
Attachment Q-Set | 12 months post-partum
  Quality of infant attachment to father
Infant-Toddler Social and Emotional Assessment (ITSEA) | 12 months post-partum
  Behavioral problems and competencies in infants

SECONDARY OUTCOMES:
Maternal depressive symptoms (Beck Depression Inventory) | 12 months post-partum
  Depressive symptoms reported by mothers
Descriptive In-home Survey of Chaos - Observer ReporteD (DISCORD) | 1 month post-partum
  Household chaos, observed, in families

OTHER OUTCOMES:
Paternal depressive symptoms (Beck Depression Inventory) | 12 months post-partum
  Depressive symptoms reported by fathers

CONTACTS AND LOCATIONS:
Locations (1):
- Douglas Teti, State College, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No